CLINICAL TRIAL: NCT05759481
Title: Prevention of Post-Operative Nausea and Vomiting With Propofol Infusion
Acronym: PONV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sonal Sharma, Assistant Professor, Department of Anesthesiology and Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00021935
Record Dates: First submitted 2023-02-22; First posted 2023-03-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Post-operative Nausea and Vomiting
Keywords: Post-Operative Nausea; Post-Operative Vomiting; propofol; motion sickness
MeSH Terms: conditions — Vomiting; Motion Sickness | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol (Experimental): Low-dose propofol infusion at 25 mcg/kg/min
  Interventions: Drug: Propofol
- Placebo (Placebo Comparator): Same volume of 0.9% normal saline as the study group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propofol — Propofol is administered starting at surgery induction and ending at skin closure
  Other Names: 2,6 di-isopropylphenol
  Arms: Propofol
Other: Placebo — Placebo is administered starting at surgery induction and ending at skin closure
  Arms: Placebo

SUMMARY:
The purpose of this study is to clarify whether or not a low-dose propofol infusion can effectively prevent postoperative nausea and vomiting (PONV) in patients who have a documented history of PONV and/or motion sickness.

DETAILED DESCRIPTION:
Propofol is administered as both low dose and as sole anesthetic in patients with history of PONV and/or motion sickness. But efficacy of one dose over the other is not studied. This study plans to clarify if propofol in low dose is as effective as its administration as sole anesthetic in patients with history of PONV and/or motion sickness

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing general anesthesia for elective surgery
2. Documented history of Patient's self-disclosure of PONV and/or motion sickness during pre-anesthesia discussions
3. No documented allergy/adverse reaction to propofol
4. English speaking
5. At least 18 years of age

Exclusion Criteria:

1. Any anti-nausea medication taken within 24 hours prior to surgery
2. Unable to provide consent independently
3. Allergy or adverse reaction to propofol
4. Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Nausea (urge to vomit) episodes | 24 hours
  Number of self-reported nausea episodes
Retching (labored, spasmodic, rhythmic contractions of respiratory muscles without expulsion of gastric contents) episodes | 24 hours
  Number of self-reported retching episodes
Vomiting (forceful expulsion of gastric contents) episodes | 24 hours
  Number of self-reported vomiting episodes

SECONDARY OUTCOMES:
Choice of antiemetic- Dexamethasone | 24 hours
  medication administered.
Number of times dexamethasone administered | 24 hours
  frequency of administration
Choice of antiemetic- Ondansetron | 24 hours
  medication administered.
Number of times ondansetron administered | 24 hours
  frequency of administration
Choice of antiemetic- Promethazine | 24 hours
  medication administered
Number of times promethazine administered | 24 hours
  frequency of administration
Choice of antiemetic- metoclopramide | 24 hours
  medication administered
Number of times metoclopramide administered | 24 hours
  frequency of administration
Choice of antiemetic- Prochlorperazine | 24 hours
  medication administered
Number of times prochlorperazine administered | 24 hours
  frequency of administration
Choice of antiemetic- Droperidol | 24 hours
  medication administered
Number of times droperidol administered | 24 hours
  frequency of administration
Choice of antiemetic- scopolamine | 24 hours
  medication administered
Number of times scopolamine administered | 24 hours
  frequency of administration
Choice of antiemetic-diphenhydramine | 24 hours
  medication administered
Number of times diphenhydramine administered | 24 hours
  frequency of administration

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Sharma, MD, Principal Investigator — Assistant Professor, Department of Anesthesiology and Perioperative Medicine
Locations (1):
- Penn State Health Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Keck WL, Deng E, Liu WM, Kanekar R, Lomivotrov V, Sharma S. Effect of low-dose propofol infusion with sevoflurane versus propofol-only total intravenous anesthesia on postoperative nausea and vomiting in high-risk patients: a single-blind randomized controlled clinical trial. BMC Anesthesiol. 2026 Jan 28. doi: 10.1186/s12871-026-03649-7. Online ahead of print. PMID 41593496